CLINICAL TRIAL: NCT03801850
Title: Quantitative Evaluation of the Breast's Morphological Variations During Radiotherapy: Monocentric Feasibility Study MorphoBreast3D
Brief Title: Quantitative Evaluation of the Breast's Morphological Variations During Radiotherapy: MorphoBreast3D
Acronym: MB3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-01; 2017-A02489-44 (Other: ANSM)
Record Dates: First submitted 2018-05-18; First posted 2019-01-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer Female; Adjuvant Radiotherapy
Keywords: volume variation; deformation; repositioning; dosimetric quality; 3D scan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observational cohort (Experimental)
  Interventions: Device: 3D surface scan

INTERVENTIONS:
Device: 3D surface scan — measurement of inter fractional deformations by surface scanning

SUMMARY:
Quantitative evaluation of the breast's morphological variations during radiotherapy consisting in performing three-dimensional surface acquisitions of the breast in order to study its shape and volume. Evaluation of the dosimetric impact of these variations.

ELIGIBILITY:
Inclusion Criteria:

* Women
* In situ or invasive breast carcinoma
* Treated by conservative breast surgery
* Pre-treatment with authorized chemotherapy
* Eligible for conventional breast irradiation in 25 sessions of 2 Gy with or without irradiation of the tumor bed and lymph nodes area
* Conventional 3D radiotherapy technique
* Bra cup size from A to D included
* Speaking and understanding french
* Having given written consent
* Patient with health insurance

Exclusion Criteria:

* Surgical treatment by mastectomy
* No indication for breast radiotherapy
* Local or diffuse inflammatory state of the breast at inclusion
* History of epilepsy or anticonvulsive treatment for preventive or curative purposes
* BMI> 30kg / m2
* T4 stage tumor
* Bilateral breast tumor
* Use of a ventilatory control to treat the patient
* Minor patient or major incompetent
* Patient deprived of liberty
* Patient under safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Impact of breast morphology or volume changes during the breast irradiation on the total dose administered | Change of the dose delivered in the breast from the baseline treatment planification at the end of the treatment (at 5 weeks for in-situ carcinoma and at 6.5 weeks for invasive carcinoma)
  To analyse the effect of morphological changes in the breast during breast radiotherapy on the dose really administered in the remaining mammary gland after breast-conserving surgery compared to the dose initially planned.

SECONDARY OUTCOMES:
Preliminary quantitative assessment of breast volume changes (mL) during breast radiotherapy following breast cancer conservative surgery | At 1, 5, 12, 19, 26, 33 and 43 days from the start of the treatment (corresponding to the fraction number 1, 5, 10, 15, 20, 25, 33)
Preliminary quantitative assessment of breast deformations (mm) during breast radiotherapy following breast cancer conservative surgery | At 1, 5, 12, 19, 26, 33 and 43 days from the start of the treatment (corresponding to the fraction number 1, 5, 10, 15, 20, 25, 33)
Breast deformation and volume measurements reproducibility | before treatment start
  Evaluation of the reproducibility of deformation and volume measurements between 2 consecutive surface scan acquisition. Reproducibility was calculated in accordance with International Organization of Standardisation (ISO 5725-2) and American Society for Testing and Material E177
Deviation between the breast volume calculated and the breast volume manually delineated | before treatment start
  Evaluation of the difference between the initial breast volume calculated by the software developed for the study and the delineated volume
Required measurement time (surface scan) | At 1, 5, 12, 19, 26, 33 and 43 days from the start of the treatment (corresponding to the fraction number 1, 5, 10, 15, 20, 25, 33)
  Mean time (in minutes) needed to perform a surface scan
Correlation between textural data and radio-induced erythema | At 1, 5, 12, 19, 26, 33 and 43 days from the start of the treatment (corresponding to the fraction number 1, 5, 10, 15, 20, 25, 33)
Potential dose distribution alteration despite no variation of the 95Recalculated or the D2Recalculated | at the end of each treatment (at 5 weeks for in-situ carcinoma and at 6.5 weeks for invasive carcinoma)

CONTACTS AND LOCATIONS:
Overall Officials: Georges NOEL, MD PhD, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre paul Strauss, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided